CLINICAL TRIAL: NCT00005939
Title: Phase I/II Study of Interstitial Colloidal 32P for Locally Recurrent Prostate Cancer Failing Radiation
Brief Title: Brachytherapy in Treating Patients With Recurrent Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Molecular Medicine (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067749; CMM-99025; NCI-V00-1585
Record Dates: First submitted 2000-07-05; First posted 2004-05-26 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2001-02

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Phosphorus-32

INTERVENTIONS:
Radiation: brachytherapy
Radiation: phosphorus P32

SUMMARY:
RATIONALE: Radiation therapy uses high-energy radiation to damage tumor cells. Brachytherapy uses radioactive material that is placed directly into or near the tumor. Brachytherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of brachytherapy in treating patients who have recurrent prostate cancer that has not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dosimetry and toxicity of interstitial colloidal phosphorus P32 (cP32) in patients with locally recurrent prostate cancer that has failed conventional therapy. II. Determine the maximum tolerated dose of interstitial cP32 when combined with interstitial macroaggregated albumin (infusional brachytherapy) in these patients. III. Determine the therapeutic response rate to acceptable single doses of cP32 in these patients.

OUTLINE: This is a dose escalation study of colloidal phosphorus P32 (cP32). Patients receive cP32 and macroaggregated albumin via interstitial infusion using ultrasound localization. Cohorts of 3 patients receive escalating doses of cP32 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 4 patients experience dose limiting toxicities. Additional patients are treated at the MTD. Patients are followed at 1, 2, 4, and 6 weeks; then at 2, 4, 8, 12, 16, 20, and 24 months; and then every 6 months thereafter until death.

PROJECTED ACCRUAL: A total of 20-25 patients will be accrued for phase I of the study and a total of 40 patients will be accrued for phase II of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locally recurrent prostate cancer that has failed conventional therapy (i.e., external beam radiotherapy, radioactive seed implants, and hormonal therapy) Must be confirmed clinically with elevated PSA and/or ultrasound Prostates between 2-5 cm in diameter (i.e., volumes of 4-65 cm3) preferred Prostates greater than 5 cm allowed, but 2 needles required for good distribution of study drug No clinical/radiographic evidence of metastatic disease No history of injury to urethra, bladder, or rectum

PATIENT CHARACTERISTICS: Age: 21 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Neutrophil count at least 1,900/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL (transfusion allowed) Hepatic: Not specified Renal: Blood urea nitrogen no greater than 25 mg/dL Creatinine no greater than 1.5 mg/dL

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics Surgery: Not specified

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Wayne S. Court, MD, PhD, Study Chair — Center for Molecular Medicine
Locations (1):
- Center for Molecular Medicine, Garden City, New York, United States